CLINICAL TRIAL: NCT05863611
Title: The Effect of Frailty on Balance and Fall Risk in Patients With Type 2 Diabetes
Brief Title: The Impact of Frailty in Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Gulsah Turanoglu, Principal Investigator, Kırıkkale University
Other Study IDs: KirikkaleUniversity711
Record Dates: First submitted 2023-01-11; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 25 individuals with frailty syndrome with type 2 diabetes
  Interventions: Other: arms
- 25 individuals without frailty syndrome with type 2 diabetes
  Interventions: Other: arms

INTERVENTIONS:
Other: arms — During the research, a questionnaire form (age, gender, educational status, etc.) in which your demographic information will be recorded for evaluation purposes and a consent form for participation in the study will be filled. Standardized Mini Mental Test will be applied. Then fragility will be evaluated with the Fried Fragility Index. Fall assessment will be assessed with the Fall Risk Self-Assessment Scale. Balance assessment will be made with the Tinetti Balance and Gait Assessment.

SUMMARY:
The purpose of our work; To investigate the effect of frailty on balance and fall risk in individuals with type 2 diabetes.The reason why participants the investigators invited to the study is participants diagnosis of Type 2 Diabetes.During the research, a questionnaire form (age, gender, educational status, etc.) in which participants demographic information will be recorded for evaluation purposes and a consent form for participation in the study will be filled. Standardized Mini Mental Test will be applied. Then fragility will be evaluated with the Fried Fragility Index. Fall assessment will be assessed with the Fall Risk Self-Assessment Scale and balance assessment will be made with the Tinetti Balance. participants will not need to spend a long time for all assessments. The time required for the assessment will be around 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes
* Being 65 years or older
* Not having a cooperation problem,
* No communication difficulties or problems voluntarily accepting participation in the research

Exclusion Criteria:

* - Those with uncontrollable hypertension, heart disease, cardiac arrhythmia
* Those with cardiovascular disease
* Those who have malignancy and cause malignancy, chemotherapy, radiotherapy
* Those with any neurological or orthopedic disorders
* Those who have had an operation in the last 6 months
* Those on bed rest
* Individuals addicted to alcohol and drugs
* Those who do not agree to participate in the research

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: be diagnosed with type 2 diabetes be over 65 years old
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2023-05-25 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
Frailty has an effect on balance in patients with type 2 diabetes. | march 15, 2023 - june 10 , 2023
  Balance assessment will be made with the Tinetti Balance

SECONDARY OUTCOMES:
Frailty has an effect on the risk of falling in patients with type 2 diabetes. | march 15, 2023 - june 10 , 2023
  Fall assessment will be assessed with the Fall Risk Self-Assessment Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Gulsah Turanoglu, Kırıkkale, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: march 15,2023 - june 10,2023